CLINICAL TRIAL: NCT02361190
Title: Effects of Fast Acting Testosterone Nasal Spray on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robert Josephs, Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014-07-0062
Record Dates: First submitted 2014-11-20; First posted 2015-02-11 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Testosterone; Testosterone Propionate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo nasal spray (Placebo Comparator): Subjects will inhale approximately 40ml aqueous solution via intranasal route
  Interventions: Drug: Placebo
- Testosterone nasal spray (Experimental): Subjects will inhale approximately 40ml aqueous, testosterone-containing solution via intranasal route
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Administration of 1ml aqueous nasal spray containing 7mg testosterone propionate
  Other Names: Testosterone propionate
  Arms: Testosterone nasal spray
Drug: Placebo — Administration of 1ml aqueous saline spray
  Other Names: saline
  Arms: Placebo nasal spray

SUMMARY:
The proposed study will test the effects of a fast-acting testosterone nasal spray on the fear reactions of young men to two distinct anxiety challenges (social and nonsocial) using a double-blind randomized experimental design.

DETAILED DESCRIPTION:
Aim 1: Test the hypothesis that men administered testosterone nasal spray will result in lower levels of anxiety (anticipatory and situational) and greater levels of approach behavior in response to two distinct (social and nonsocial) anxiety challenges relative to men administered placebo spray.

Aim 2: Test the hypothesis that anxiety challenge type (social versus nonsocial) will moderate the effects of testosterone administration on subjects' responses to challenge.

Aim 3: Test the hypothesis that rejection sensitivity - heightened sensitivity to evaluative threat - will moderate the effects of drug condition on response to the two anxiety challenge tests.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 years of age or older

Exclusion Criteria:

* Male breast cancer
* Obstructive sleep apnea
* Suspected or diagnosed prostate cancer
* Male breast cancer
* Obstructive sleep apnea
* Diabetes
* Heart Disease
* Liver disease (e.g., hepatitis)
* Kidney disease
* Thyroid disease
* Tuberculosis or history if positive TB test
* Infection or fever in the past 7 days
* Surgeries within the last 6 weeks
* Anemia
* Gastrointestinal disease
* Respiratory disease (e.g., asthma or chronic bronchitis)
* Other (Please list)
* Reynaud's Disease
* Type 2 diabetes
* Diagnosed hypersensitivity to cold
* Warfarin (Coumadin) for thinning blood
* Insulin or any oral drugs for diabetes
* Propranolol (Inderal)
* Oxyphenbutazone
* Imipramine
* Any kind of corticosteroid drug
* Insulin
* Steroids
* Statins (i.e.., cholesterol lowering drugs)
* Sleeping pills
* Drugs to treat hormone disorders
* Antibiotics in the past 7 days
* Gastrointestinal disease
* Pain Killers -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Magnitude of behavioral approach | 30 minutes
  Subjects will be asked to approach a fearful object. Approach will be measured as number of steps (out of 18) the subject completes, with each step bringing the subject closer to the target object

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Josephs, Phd, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin Department of Psychology, Austin, Texas, United States